CLINICAL TRIAL: NCT04032483
Title: A Survey of Financial Toxicity of Radiation Treatment in Rural Cancer Patients
Brief Title: A Survey of Financial Toxicity in Rural Cancer Patients
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nirav.S.Kapadia, Principal Investigator, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19068
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Financial Toxicity
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to elucidate the prevalence of financial toxicity, identify significant risk factors for toxicity, and understand the burdens of the specific St. Johnsbury rural population. These data will drive future, larger studies to investigate how to alleviate the burden of financial toxicity, especially in vulnerable patient populations.

DETAILED DESCRIPTION:
"Financial toxicity" refers to a side effect of cancer treatment that is financial in nature, and has become increasingly important to oncologists, patients, and researchers because of its implications in adverse social outcomes for patients. Financial toxicity in the context of cancer care is the monetary cost, and subsequent social implications of the cost, on patients undergoing cancer treatment. Although financial toxicity for patients undergoing cancer treatment has some research attention, financial toxicity associated with radiation therapy for cancer patients has not. There is preliminary data that has shown that there are two forms of financial toxicity: the direct cost of cancer therapy (medical services) and the indirect costs (gas for travel, lost wages for sick days, etc.). However, the degree of cost and sources have not been fully investigated. Specifically, financial toxicity in the context of cancer patients from rural populations (such as those at NCCC) has not been fully explored. This project will attempt to understand the salient factors, costs, and magnitudes of financial toxicity in radiation therapy that will allow for more targeted studies to investigate vulnerable patient populations who experience greater financial toxicity.

Study recruitment temporarily halted due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing treatment at Norris Cotton Cancer Center North, St. Johnsbury, VT
* Current radiation/oncology patient
* Ability to speak or write in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: With 100 participants, we are trying to show the prevalence of financial toxicity in radiation patients and make our findings as generalizable as possible to the broader population of rural radiation oncology patients in the US.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Financial toxicity | The time frame will once a week for 3-9 weeks, dependent on the treatment duration of the patient.
  Both qualitative and quantitative surveys will be given to patients and will ask them for their financial information. These surveys will be given each week, on the day the physician sees the patient. The survey will ask for the following information to determine their direct costs of radiation treatment: employment, race, ethnicity, gender, income, insurance status, co-payments, wage-earner status, out-of-pocket costs for treatment, transportation to treatments, and drug costs. The survey will also ask questions to determine their indirect costs of radiation treatment: productivity days lost, disability days, if they have sold anything in the past week, if they have cut down on leisure activities, concern about paying for bills, ability to meet monthly expenses, and how much they deem their cancer treatment has impacted their satisfaction with financial status.

CONTACTS AND LOCATIONS:
Locations (1):
- Norris Cotton Cancer Center, Saint Johnsbury, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided